CLINICAL TRIAL: NCT07137650
Title: A Game-based Screening for Mild Cognitive Impairment Detection in Older Adults
Brief Title: A Game-based Screening for MCI Detection in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00142237
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research explores a new and engaging way to screen for mild cognitive impairment (MCI) in older adults using a computer game instead of traditional paper-based tests. MCI is an early sign of cognitive decline and can lead to dementia. Detecting it early is important, but current methods are not always accessible, enjoyable, or reflective of real-life tasks.

The study will test the Glenrose Grocery Game (G3), a computer game simulating a real-life shopping trip. The game challenges memory, attention, and problem-solving in a familiar, interactive setting. Originally developed for cognitive training in older adults, this is the first time it is being tested as a screening tool for cognitive issues.

Fifty-nine older adults (aged 65+) will be recruited, with and without signs of MCI. Each participant will attend a single 90-minute session. They will provide consent, complete demographic questions, and undergo two standard cognitive tests: the Montreal Cognitive Assessment (MoCA) and Quick Mild Cognitive Impairment screen (Qmci). Anxiety will be measured before and after the cognitive tasks. Participants will then play six levels of the G3 game and complete a usability questionnaire.

The study will measure game performance (e.g., time taken, errors, and budget management), cognitive test scores, anxiety levels before and after gameplay, and usability ratings.

The G3 game could provide a less stressful, more realistic, and more accessible method to screen for memory problems, potentially enabling earlier detection. It may be especially helpful for people with limited access to trained clinicians or those who feel anxious during traditional tests. Risks are minimal, similar to daily activities, such as feeling tired or briefly anxious. Participants may stop at any time. All data will be kept private and secure, with names replaced by ID numbers.

DETAILED DESCRIPTION:
Eligibility: Adults aged 65+ with typical cognition or mild concerns, with adequate vision, hearing, and ability to use a mouse, and able to understand English and give consent.

Locations: Community centres, long-term care homes, the University of Alberta, or participants' homes.

Recruitment: Social media, posters, word of mouth, and community presentations. Benefits: No direct benefit, but participants may enjoy the game and contribute to testing a potentially more user-friendly screening method for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults who are aged 65 and above with typical cognition or MCI as reported by themselves, or a health care professional.
* Older adults participating in this study must have MoCA score of 18 or higher.
* Older adults participating in the study must have functional vision and hearing, with or without aids such as glasses or hearing aids that enable them to interact with the game and comprehend the instructions. As part of the study recruitment activities, the researcher will explain the tasks required and discuss the vision and hearing demands.
* Older adults participating in the study must be capable of communicating and comprehending assessments, instructions, and simple sentences in English, as communication and comprehension is essential for interacting effectively with game components and the researcher. To assess their communication, reading, and comprehension skills, the researcher will provide participants with a few sentences in English related to the game content. Participants will be asked to read these sentences aloud and explain the meaning of the sentence to confirm their ability to read and understand the content.
* Older adults participating in the study must have adequate upper extremity function to play the game, using a mouse and do paper-and-pencil based measurements, using a pencil. During the study's introduction and training part of the game, potential participants can report any physical limitations. The researcher will also screen for these

Exclusion Criteria:

• Older adults currently suffering from Influenza, COVID-19, or any other viral illness at the time of data collection that could impair their performance will be excluded. These conditions could impair their performance, potentially affecting the reliability of the outcomes. Additionally, the presence of such illnesses could pose a health risk to other participants who use the same equipment, as well as to the researcher.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults who are 65 and older with and without mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
1. Montreal Cognitive Assessment (MoCA) | Time Frame: Administered once during the 90-minute session. The administration of this test takes 10-15 minutes
  1. A standard cognitive screening tool to assess general cognitive abilities. Range: 0-30 interpretation: Higher scores indicate better cognitive performance.
  2. A brief screening test to detect early cognitive impairment.
  3. Task completion, Time of playing, Number of correct and errors, using aid,..
  4. System usability scale to measure the participants' experience with the game
  5. State and train anxiety of the participants
Quick Mild Cognitive Impairment screen (Qmci) | Time Frame: Administered once during the 90-minute session.The administration of this test takes 10-15 minutes
  Description: A brief screening instrument for early detection of mild cognitive impairment.
  Range: 0-100 points. Range: 0-100 points.
  Interpretation: Higher scores indicate better cognitive performance. Interpretation: Higher scores indicate better cognitive performance.
Game Performance Measures from the Glenrose Grocery Game (G3) | Time Frame: Collected continuously during gameplay within the 90-minute session. Gameplay usually takes 30 minutes.
  Description: Objective in-game performance metrics including task completion status, total play time, number of correct responses, number of errors, and use of in-game aids. Score Range: Variable depending on the specific metric (e.g., errors = 0 to maximum possible errors per stage).
  Interpretation: Higher accuracy and fewer errors indicate better cognitive performance.

SECONDARY OUTCOMES:
System Usability Scale (SUS) System Usability Scale (SUS) System Usability Scale (SUS) | Time Frame: Administered immediately after gameplay during the same 90-minute session. It takes 5 minutes to do this self-adminstred test.
  Description: A validated 10-item questionnaire assessing participants' perceived usability of the G3 game.
  Score Range: 0-100 points.
  Interpretation: Higher scores indicate better usability.
State-Trait Anxiety Inventory (STAI) | Time Frame: Administered before and after gameplay during the same 90-minute session. Doin the test takes aorund 15 minutes
  Description: A standardized measure of participants' temporary (state) and general (trait) anxiety levels.
  Score Range: 20-80 points for each subscale.
  Interpretation: Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Rios Rincon, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zygouris S, Iliadou P, Lazarou E, Giakoumis D, Votis K, Alexiadis A, Triantafyllidis A, Segkouli S, Tzovaras D, Tsiatsos T, Papagianopoulos S, Tsolaki M. Detection of Mild Cognitive Impairment in an At-Risk Group of Older Adults: Can a Novel Self-Administered Serious Game-Based Screening Test Improve Diagnostic Accuracy? J Alzheimers Dis. 2020;78(1):405-412. doi: 10.3233/JAD-200880. PMID 32986676

DOCUMENTS (1):
  • Study Protocol (2024-08-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT07137650/Prot_000.pdf